CLINICAL TRIAL: NCT04428138
Title: Observational Cross-sectional Study on the Association Between Inguinal Hernias and Arterial Diseases
Brief Title: Inguinal Hernia and Arterial Disease
Acronym: HEARD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Other Study IDs: ER.ALL.2018.30
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Inguinal Hernia; Arterial Disease
Keywords: Inguinal Hernia; Arterial Disease; Peripheral artery disease; Carotid stenosis; Arterial aneurysm
MeSH Terms: conditions — Hernia, Inguinal; Peripheral Arterial Disease; Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Inguinal hernia: Patients presenting with inguinal hernia will undergo vascular in-office visit and echo duplex of aorta, carotid arteries and lower limb arteries in order to detect any abnormalities related to arterial disease (aneurysm, stenosis, flow alteration).
  Interventions: Diagnostic Test: In-office vascular visit; Diagnostic Test: Echo duplex scan of arterial system

INTERVENTIONS:
Diagnostic Test: In-office vascular visit — Every patient will undergo a complete physical examination in order to detect any clinical or sub clinical vascular disease.
Diagnostic Test: Echo duplex scan of arterial system — Every patient will undergo a complete echo duplex scan in order to detect any morphological or hemodynamic alteration of aorta, carotid arteries and lower limb arteries.

SUMMARY:
Inguinal hernias are associated with problems related to the venous system by the linking to extracellular matrix alterations (ECM). On the other hand, arterial diseases (arterial aneurysms, carotid, stenosis, peripheral artery disease) are widespread in the general population and may share others pathological pathways related to ECM impairment. Aim to this study is to evaluate the prevalence of arterial diseases in patients with inguinal hernia.

DETAILED DESCRIPTION:
Previous studies showed the correlation between inguinal hernias and venous disease. The common pathophysiological pathway between these clinical conditions is linked to extracellular matrix (ECM) alterations. Arterial diseases, mainly represented by carotid stenosis, peripheral artery disease and arterial aneurysms, are widespread in western population and are responsible of high rates of morbidity and mortality. These diseases are also related to some ECM alterations.

Aim of this cross-sectional study is to evaluate the prevalence of arterial disease among patients with inguinal hernias. The primary endpoint of this study is to provide new epidemiological evidences on this association that may help physicians in novel preventive strategies. The study will consider the inclusion of consecutive patients assessed for inguinal hernia over 1 year period in order to study the prevalence of concomitant arterial disease, by means of office visit, echo duplex scan of the aorta and its main branches, carotid arteries and lower limb arteries.

ELIGIBILITY:
Inclusion Criteria:

* patients with inguinal hernia

Exclusion Criteria:

* patients with malignancies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of the general population presenting with inguinale hernia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of arterial disease in patients with inguinal hernia | at 1 year
  Patients with inguinal hernia will be assessed for the presence of arterial aneurysm, carotid stenosis, and peripheral artery disease in order to find any correlation between these pathological conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Serra, M.D., Ph.D., Principal Investigator — University Magna Graecia of Catanzaro
Locations (2):
- Italy (2):
  - CIFL- Interuniversity Center of Phlebolymphology, Catanzaro
  - University Magna Graecia of Catanzaro, Catanzaro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serra R, Buffone G, Costanzo G, Montemurro R, Scarcello E, Stillitano DM, Damiano R, de Franciscis S. Altered metalloproteinase-9 expression as least common denominator between varicocele, inguinal hernia, and chronic venous disorders. Ann Vasc Surg. 2014 Apr;28(3):705-9. doi: 10.1016/j.avsg.2013.07.026. Epub 2013 Oct 31. PMID 24184457
- [Background] Serra R, Buffone G, Costanzo G, Montemurro R, Perri P, Damiano R, de Franciscis S. Varicocele in younger as risk factor for inguinal hernia and for chronic venous disease in older: preliminary results of a prospective cohort study. Ann Vasc Surg. 2013 Apr;27(3):329-31. doi: 10.1016/j.avsg.2012.03.016. Epub 2012 Sep 19. PMID 22998788
- [Background] Rowse PG, Crestanello JA. Commentary: Abdominal wall hernia: An important risk association in aortic aneurysmal disease or just a dull ache? J Thorac Cardiovasc Surg. 2021 Dec;162(6):1678-1679. doi: 10.1016/j.jtcvs.2020.03.105. Epub 2020 Apr 6. No abstract available. PMID 32448686